CLINICAL TRIAL: NCT03935399
Title: Effects of Intramuscular Oxytocin on Sensory Function in Healthy Volunteers With Ultraviolet Burn Injury to the Skin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00056660
Record Dates: First submitted 2019-04-24; First posted 2019-05-02 (Actual); Results first posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Double blinded crossover treatment with oxytocin and placebo (saline)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant, Investigator and outcomes assessor will be blinded. Research Pharmacist will prepare the study medication administration and hold the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oxytocin first, then saline placebo (Other): Intramuscular injection of oxytocin (Pitocin®), 10 IU on the first study day and of 1 ml saline placebo on the second study day
  Interventions: Drug: Oxytocin; Drug: Saline
- Saline placebo first, then oxytocin (Placebo Comparator): Intramuscular injection of 1 ml saline placebo on the second study day and of oxytocin (Pitocin®), 10 IU on the second study day
  Interventions: Drug: Oxytocin; Drug: Saline

INTERVENTIONS:
Drug: Oxytocin — 10 IU oxytocin (Pitocin) for intramuscular injection
  Other Names: Pitocin
Drug: Saline — 1.5 ml preservative free saline for intramuscular injection

SUMMARY:
This study proposes to evaluate the effects that a dose of oxytocin given by intramuscular (IM) injection (into the muscle) will have on an area of skin that has been exposed to ultraviolet (UV) light. The area of skin exposed to UV light will have a mild sun burn feeling.

Sensory testing will be performed on the area of UV burn. The area will be evaluated for sensitivity in 3 methods: touch, vibratory

DETAILED DESCRIPTION:
This protocol aims to provide an estimate of effect size of intramuscular oxytocin on a test of Aβ and of Aδ fiber sensitivity in injured skin following ultraviolet B (UVB) burned skin.

For the primary goal - to examine the effects of oxytocin peripheral nerves after tissue injury - the investigators chose the controlled ultraviolet sunburn model.

The investigators propose a randomized, blinded, cross over design with treatment with oxytocin one day and placebo on another. Following baseline measures on each of the two study days, participants will receive an intramuscular injection of oxytocin (Pitocin®) in its indicated dose of 10 IU (17 μg) or an equivalent volume of saline.

In order to determine the highest frequency that Aβ nerve fibers can respond to, the investigators will use a device that produces an oscillatory / vibratory stimulus which can be used on the hand.

Pain threshold to punctate stimulation within the area of irradiation will be determined using calibrated von Frey filaments and an up-down sequential method which efficiently estimates median thresholds.

Thermal heat testing will also be performed by the surface of the skin of the forearm or leg is heated to 45°C using a computer controlled thermode for a period of 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 18 and < 60 years of age,
* Body Mass Index (BMI) <40
* Generally in good health as determined by the Principal Investigator based on prior medical history
* Normal blood pressure and resting heart rate without medication

Exclusion Criteria:

* Hypersensitivity, allergy, or significant reaction to any ingredient of Pitocin®
* Any disease, diagnosis, or condition (medical or surgical) that, in the opinion of the Principal Investigator, would place the subject at increased risk
* Women who are pregnant (positive result for serum pregnancy test at screening visit), women who are currently nursing or lactating, women that have been pregnant within 2 years.
* Neuropathy, chronic pain, diabetes mellitus, or taking benzodiazepines or pain medications on a daily basis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C Eisenach, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: First Study Day
Arm/Group | Oxytocin First, Then Saline Placebo | Saline Placebo First, Then Oxytocin
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Second Study Day
Arm/Group | Oxytocin First, Then Saline Placebo | Saline Placebo First, Then Oxytocin
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin First, Then Saline Placebo | Saline Placebo First, Then Oxytocin | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (12) | 40 (12) | 38 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29 (5) | 26 (3) | 27 (4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Vibration Frequency Detection Threshold (When Vibration is First Felt) After IM Injection
Description: Vibration frequency detection threshold in the burned area after IM Oxytocin or placebo injection will be obtained by the subject placing the forearm area that was exposed to the UV burn on the oscillatory device and informing the investigators when the first perception of vibration is felt. A recording of the frequency (1 kilo Hertz to 1 Hertz) will be documented.
Time Frame: From 5 minutes to 120 minutes
Population: Please note that the protocol was amended after the first 5 participants. The first 5 participants were tested for vibration FREQUENCY detection threshold and the last 5 participants were tested for vibration INTENSITY detection threshold. This outcome relates to the first 5 participants only.
Measure: Mean (Standard Deviation); unit: Hz
Groups:
- Placebo: Saline: 1.5 ml preservative free saline for intramuscular injection
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 5 | 5
Hz | 22 (14) | 21 (8)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Exploratory analysis without power calculation; Test type: Superiority — Exploratory analysis without power calculation; p = 0.83, ANOVA; Repeated measures one factor ANOVA

2. Primary Outcome: Change in Pain Threshold (the Point Where Pain is First Perceived) to a Punctate Mechanical Stimulus After IM Injection.
Description: Verbal pain punctate stimulus detection threshold (the point where pain is first perceived) in the burned area after IM Oxytocin or Placebo injection will be obtained by using von Frey filaments (small filaments that are similar to a paint brush bristle). The skin will be touched with the filaments and the participant will state when pain is perceived and the size of the filament will be documented.
Time Frame: From 5 minutes to 120 minutes
Population: Please note that the protocol was amended after the first 5 participants. The first 5 participants were tested for pain THRESHOLD to mechanical stimulation and the last 5 participants were tested for degree of pain INTENSITY to a fixed mechanical stimulation. This outcome relates to the first 5 participants only.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 5 | 5
grams | 0.20 (0.66) | 0.29 (0.55)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Exploratory analysis without power calculation; Test type: Superiority — Exploratory analysis without power calculation; p = 0.92, ANOVA; One factor repeated measures ANOVA

3. Primary Outcome: Change in Hypersensitivity to Von Frey Filament (225 milliNewton) After IM Injection.
Description: Hypersensitivity in the burned area after IM Oxytocin or placebo injection will be obtained by using a von Frey filament (small filament that is similar to a paint brush bristle). The skin will be touched with the filament and the participant will state when sensitivity is perceived and the area marked and measured in centimeters squared.
Time Frame: From 5 minutes to 65 minutes
Population: Please note that the protocol was amended after the first 5 participants. The first 5 participants were tested for pain THRESHOLD to mechanical stimulation and the last 5 participants were tested for degree of pain INTENSITY to a fixed mechanical stimulation. This outcome relates to the last 5 participants only.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 5 | 5
cm^2 | 6.4 (8.6) | 8.8 (8.6)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Exploratory analysis without power calculation; Test type: Superiority — Exploratory analysis without power calculation; p = 0.79, ANOVA; One factor repeated measures ANOVA

4. Primary Outcome: Change in Vibration Frequency Detection of Fixed Frequency (When Vibration is First Felt) After IM Injection
Description: Vibration frequency detection of a fixed frequency (256 Hertz) in the burned area after IM Oxytocin or placebo injection will be obtained. The subject will place the wrist area that was exposed to the UV burn on the oscillatory device, the fixed vibratory frequency will begin and will be increased in intensity and the subject will inform the investigators when the first perception of vibration is felt. A recording of the intensity level will be documented in Hertz.
Time Frame: From 5 minutes to 65 minutes
Population: Please note that the protocol was amended after the first 5 participants. The first 5 participants were tested for vibration FREQUENCY detection threshold and the last 5 participants were tested for vibration INTENSITY detection threshold. This outcome relates to the last 5 participants only.
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 5 | 5
Hz | 1.8 (1.4) | 1.7 (3.9)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Test type: Superiority — Exploratory analysis without power calculation; p = 0.93, ANOVA — Exploratory analysis without power calculation; One factor repeated measures ANOVA

5. Secondary Outcome: Change in Sustained Heat After IM Injection Non Dominant Arm
Description: Verbal pain scores (0 to 10; 0 is equivalent to no pain and 10 is equivalent to the worst pain imaginable) to 45 degree Celsius temperature after IM Oxytocin or placebo injection.
Time Frame: From 21 minutes to 125 minutes
Population: Please note that the protocol was amended after the first 5 participants. The first 5 participants were tested for pain report to sustained heat applied to the ARM and the last 5 participants were tested for pain report to sustained heat applied to the LEG. This outcome relates to the first 5 participants only.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale | -0.30 (0.65) | -0.70 (0.84)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Test type: Superiority — Exploratory analysis without power calculation; p = 0.89, ANOVA — Exploratory analysis without power calculation; Two factor repeated measures ANOVA

6. Secondary Outcome: Change in Sustained Heat After IM Injection
Description: Verbal pain scores (0 to 10; 0 is equivalent to no pain and 10 is equivalent to the worst pain imaginable) to 40 degree Celsius temperature applied to the site of the UV burn after IM Oxytocin or placebo injection.
Time Frame: From 36 minutes to 40 minutes
Population: Please note that the protocol was amended after the first 5 participants. Only the last 5 participants were tested for pain report to sustain heat applied at the site of the UV-B burn.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 5 | 5
score on a scale | 0.10 (0.22) | -0.20 (0.45)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Test type: Superiority — Exploratory analysis without power calculation; p = 0.83, ANOVA — Exploratory analysis without power calculation; Two way repeated measures ANOVA

7. Secondary Outcome: Change in Sustained Heat After IM Oxytocin or Placebo Injection (Lower Leg)
Description: Verbal pain scores (0 to 10; 0 is equivalent to no pain and 10 is equivalent to the worst pain imaginable) to 45 degree Celsius temperature applied to the calf (lower leg) after IM Oxytocin or placebo injection.
Time Frame: From 21 minutes to 65 minutes
Population: Please note that the protocol was amended after the first 5 participants. The first 5 participants were tested for pain report to sustained heat applied to the ARM and the last 5 participants were tested for pain report to sustained heat applied to the LEG. This outcome relates to the last 5 participants only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 5 | 5
score on a scale | -0.55 (0.94) | 0.10 (0.55)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Test type: Superiority — Exploratory analysis without power caclulation; p = 0.57, ANOVA — Exploratory analysis without power caclulation; Two way repeated measures ANOVA

ADVERSE EVENTS:
Time Frame: 5 Days
Description: This is a randomized, blinded, cross over design with treatment with oxytocin one day and placebo on another. Following baseline measures on each of the two study days, participants received an intramuscular injection of oxytocin (Pitocin®) in its indicated dose of 10 IU (17 μg) or an equivalent volume of saline.
Arm/Group | Oxytocin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/99/NCT03935399/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-10-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT03935399/Prot_SAP_001.pdf